CLINICAL TRIAL: NCT05844683
Title: Effect Of Bath Wıth Chlorexıdıne On Protectıon Of Skın Integrıty And Preventıon Of Hospıtal Infectıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, zühal çavuşoğlu, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1282
Record Dates: First submitted 2023-01-23; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Health Care Associated Infection; Skin
Keywords: skin integrity; health care associated infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Bath (Experimental): All patients in the randomized to the intervention arm will receive baths using a 2% chlorhexidine digluconate solution
  Interventions: Other: 2% chlorhexidine digluconate solution
- usual bath (Active Comparator): All patients in the randomized to the intervention arm will receive baths using soap and water according to the current practice
  Interventions: Other: usual baths

INTERVENTIONS:
Other: 2% chlorhexidine digluconate solution — Bathing will be performed at least daily using 2% chlorhexidine digluconate solution with surface-active agents on all applicable bathing surfaces, which consists of the entire body surface of the patient except eyes, inner ear, oral mucosa, and areas of loss of skin continuity (such as burnt areas, pressure injuries, etc.)
  Other Names: chlorhexidine baths
  Arms: Chlorhexidine Bath
Other: usual baths — Bathing will be performed at least daily using shampoo and water (performed according to the current practice in each center) on all applicable bathing surfaces, which consists of the entire body surface of the patient except eyes, inner ear, oral mucosa, and areas of loss of skin continuity (such as burnt areas, pressure injuries, etc.)
  Other Names: shampoo and water baths
  Arms: usual bath

SUMMARY:
The study was designed in a randomized controlled experimental design type to determine the effect of a 2% chlorhexidine bath applied in the pediatric intensive care unit on protecting skin integrity and preventing hospital-acquired infection. Research data were collected from pediatric patients aged 2 months to 18 years old, who were treated in the Pediatric Intensive Care Unit of a tertiary education and research hospital between September 2022 and September 2023. In data collection; "Child Follow-up Form", "Skin Integrity and Nosocomial Infection Follow-up Form", and "Northampton Pediatric Skin Evaluation Scale (CCRS)" were used. The data were evaluated with appropriate statistical methods in SPSS (Statistical Package for Social Sciences) for Windows 24.0 package program.

DETAILED DESCRIPTION:
The study is planned to be carried out between September 2022 and September 2023 in the 15-bed pediatric intensive care unit of Sarıyer Hamidiye Etfal Hospital. Sample size was determined by power analysis. Based on the percentage measurement values of the methods to be studied in the literature review, the total sample size was found to be n=68, with an effect size of 0.8 (cohen), a power of 90%, and a margin of error of 0.05, using the G-POWER program. The sample of the study was determined as 68 children, 34 of whom were bathed with 2% Chlorhexidine soap and 34 children who were bathed with water and soap. The randomization of the groups will be determined by drawing lots.

The pediatric intensive care unit works in two shifts, 08-17 and 16-08. During the research, the researcher will be in the clinic during the procedure, bathroom applications will be made by the research nurse in the 08-17 shift and recorded in the data collection form. A blood culture will be taken at the first hospitalization for each child who meets the acceptance and exclusion criteria of the study hospitalized in the pediatric intensive care unit, and their names will be written on closed papers by randomization drawing method and randomly thrown into the lanterns representing the control and intervention groups prepared beforehand. process will be started. Those with negative culture results at their first admission to the clinic will be included in the study.

It is known that healthcare-associated infections occur within 48 to 72 hours of hospitalization. For this reason, for both groups included in the study, necessary blood tests and cultures will be taken at their first admission to the clinic in order to evaluate the effects of the products to be used in the care process on health care-associated infections. During the application, children will be monitored daily by suspecting any systemic inflammatory response syndrome (such as fever, vomiting, diarrhea) in terms of healthcare-associated infections, and in case of any symptoms, their examinations will be repeated and recorded in the data collection form.

For the control and intervention groups, daily bathing will be done during the patient's stay in the clinic, skin evaluation will be made with the Northempton Pediatric Skin Evaluation Scale before the application, and the application process will begin for the pediatric patients whose scale score is between low and medium level and will be evaluated daily after the application. If a change is noted in the Northempton Pediatric Skin Rating Scale skin score during daily evaluations, the evaluations will continue within the intervals specified in the form of the scale, and the study will be terminated for children whose scale score is evaluated in the high-risk group. In addition, the evaluation of skin integrity will be recorded daily on the data collection form immediately after each application (dryness, redness, deterioration of skin integrity/peeling). Immediately after each application and 6 hours after the FCM-2 Skin Oil and Moisture Meter (With this device, the fat and moisture ratios of any part of the body can be determined and the measurements are concluded with high precision. Measuring range; 0%…99.9% RH) device. skin moisture values will be measured from three different regions, namely forearm, lateral upper leg and abdomen (2 cm above the umbilicus) and recorded daily in the data collection form.

Reproductive findings of healthcare-associated infections will be determined by evaluating the results of the samples sent to Sarıyer Hamidiye Etfal Training and Research Hospital laboratory.

In the study, "Northempton Pediatric Skin Evaluation Scale Turkish Version" will be used for risk assessment of skin integrity. The validity and reliability of the Turkish version of the scale was determined by Uysal et al. (2017) made by The scale is used to evaluate the skin of inpatients in pediatric clinics. Scale child's skin; weight, nutritional status, activity, bladder/bowel control, pain status, and skin condition. Each subscale consists of a total of 18 items with certain criteria. The lowest score to be obtained from the items in the scale was determined as zero and the highest score as 12. In the scale, 2 points will be added to the total score for each of the conditions such as radiotherapy, chemotherapy, steroid treatment, diabetes mellitus, staying in surgery for more than 2 hours, having a splint/cast in the body, anemia (hb: less than 8), sensory loss. A low risk of skin complications between 0-4 points in the scale and once-daily evaluation is recommended. A score of 5 to 8 is at moderate risk for skin complications, and twice-daily evaluation is recommended. It is recommended that skin complications may develop at a high risk with a score of 9 and above, and it is recommended to be evaluated every 4-6 hours or according to the situation. The higher the score on the scale, the higher the risk of skin complications in children who underwent the scale application.

The data obtained in the research is SPSS (Statistical Package for Social Analysis using the Sciences) for Windows 24.0 program will be. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. Before the data analysis, normality test will be done to test the suitability to the parametric test methods. In order to test the normal distribution condition, Kolmogorov Smirnov Z test will be applied. Chi-square and Fisher's exact tests will be applied to determine the homogeneity of the groups. In line with the results, the data will be analyzed with the related tests (Independent t-test, ANOVA, Man Whitney U, Kruskal Wallis). The findings will be evaluated at the 95% confidence interval and the significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

- • Between 2 months -18 years old,

* Receiving treatment in the pediatric intensive care unit for at least three days,
* No nosocomial infection before the first 48-72 hours of hospitalization,
* Not using antibiotics in the first hospitalization,
* Not having any skin problems,
* Evaluated as low or moderate by the Northempton pediatric skin rating scale,
* Children who were accepted to be included in the study by their parents were included in the study.

Exclusion Criteria:

* • Positive blood cultures at the first admission to the clinic,

  * Having a diagnosis and treatment that suppresses the immune system,
  * Followed up with the diagnosis of cancer,
  * Receiving steroid therapy for 10 days or more,
  * Having arterial catheterization,
  * In the postoperative period, the integrity of the skin is impaired, the operation scar,
  * Having a skin disease known to affect the skin barrier function,
  * Those with burn injuries,
  * Children with a known history of allergy to chlorhexidine were not included in the study.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
skin integrity | From admission to discharge, up to 3 days
  Northampton Pediatric Skin Assessment Tool was used for skin integrity
hospital acquired infection | From admission to discharge, up to 3 days
  incidence of hospital acquired infection

CONTACTS AND LOCATIONS:
Locations (1):
- Okan Üniversitesi, Istanbul, Turkey (Türkiye)